CLINICAL TRIAL: NCT03380507
Title: Evaluation of Hydrocortisone, Vitamin C and Thiamine for the Treatment of Septic Shock
Acronym: HYVITS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The research is no longer funded and terminated due to futility
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17207
Record Dates: First submitted 2017-12-07; First posted 2017-12-21 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2019-02

CONDITIONS: Septic Shock; Critical Illness
Keywords: Septic Shock; Vitamin C; Thiamine; Hydrocortisone; Critically Ill
MeSH Terms: conditions — Shock, Septic; Critical Illness | interventions — Hydrocortisone; Ascorbic Acid; Thiamine

STUDY DESIGN:
Intervention Model Description: Open label, prospective, randomized, two-arm parallel-group trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Triple therapy group (Experimental): Experimental group will receive usual care according to Hamad Medical Corporation Adult Sepsis Care Pathway (CPW 10311, May 2017) PLUS triple therapy.
  Triple therapy regimen:
  Intravenous vitamin C (1.5 gm q 6 hourly for 4 days or until ICU discharge, whichever is earlier), hydrocortisone (50 mg q 6 hourly for 7 days or until ICU discharge, whichever is earlier, followed by a taper over 3 days) as well as intravenous thiamine (200 mg q 12 hourly for 4 days or until ICU discharge, whichever is earlier).
  Interventions: Drug: Triple therapy group
- Control group (No Intervention): Control group will receive usual care only according to Hamad Medical Corporation Adult Sepsis Care Pathway (CPW 10311, May 2017).

INTERVENTIONS:
Drug: Triple therapy group — Refer to arms description
  Other Names: Hydrocortisone, Vitamin C and Thiamine
  Arms: Triple therapy group

SUMMARY:
Despite recent medical advances, sepsis and septic shock remain a major cause of death. Sepsis is a syndrome with a wide array of physiologic, pathologic, and biochemical abnormalities.

Several studies have shown vitamin C have decreased the circulating pro-inflammatory cytokines and oxidative stress.Thiamine had favorable effects on pro-inflammatory cytokines, oxidative stress and cellular hypoxia.The use of hydrocortisone in combination with vitamin C will increase the transport of vitamin C into the cells; since the pro inflammatory cytokines have shown to decrease the expression of the sodium-vitamin C transporter-2 (SVCT2) while glucocorticoids increase the SVCT2 expression.

A recent small retrospective study , showed a significant decrease in mortality when patients with severe sepsis and septic shock are treated with a combination of Hydrocortisone, Vitamin C, and Thiamine. Conducting a similar study with a prospective randomized design will give clinicians all over the world more answers and will help clinicians to provide better care to millions of patients using highly safe therapeutic regimen.

The objective of the current study is to explore the clinical benefits of using a combination of hydrocortisone, vitamin C, and thiamine (triple therapy) for the management of septic shock. To achieve this objective, we will compare two alternative treatment strategies, either triple therapy or usual care in patients with septic shock.

First aim: To assess the effectiveness of the triple therapy for septic shock

Second aim: To assess the safety of triple therapy

DETAILED DESCRIPTION:
Critically ill patients have low plasma levels of vitamin C. Additionally, ascorbic acid levels were inversely correlated with multi-organ dysfunction. Several studies have shown the benefit of using Vitamin C for treatment of critically ill patients; these benefits included dose dependent decrease in the SOFA score, lower vasopressor doses and duration, and lower fluid resuscitation requirements. Additionally, Intravenous Vitamin C has been shown to be safe and tolerable.

A small study demonstrated that septic shock is associated with thiamine deficiency. Additionally, a randomized controlled trial has shown that intravenous thiamine has decreased lactate levels and mortality in a subgroup of patients with thiamine deficiency. However, this benefit was not observed in the entire population of the study.

A recent study examined the effect of early treatment of patients with severe sepsis and septic shock with a combination of hydrocortisone, vitamin C, and thiamine and demonstrated a significant reduction in mortality as well as preventing organ failure progression. In this study, It has been suggested that this combination of the three agents work synergistically. The use of hydrocortisone in combination with vitamin C will increase the transport of vitamin C into the cells; since the pro inflammatory cytokines have shown to decrease the expression of the sodium-vitamin C transporter-2 (SVCT2) while glucocorticoids increase the SVCT2 expression. In an in vitro study a combination of hydrocortisone and vitamin C preserved the endothelial integrity of the lung vascular endothelial cells which was exposed to endotoxins. On the other hand either agent alone was not effective in comparison to placebo.

The objective of the current study is to explore the clinical benefits of using a combination of hydrocortisone, vitamin C, and thiamine (triple therapy) for the management of septic shock. To achieve this objective, we will compare two alternative treatment strategies, either triple therapy or usual care in patients with septic shock.

First aim: To assess the effectiveness of the triple therapy for septic shock Second aim: To assess the safety of triple therapy

1. Study Sites The study will be conducted in two hospitals (4 intensive care units) throughout the State of Qatar. All of the participating sites are part of Hamad Medical Corporation; the sites will include the MICU and SICU at Hamad General Hospital and the MICU and SICU at Al Wakra Hospital.
2. Initial screening The initial assessment will take place in the ED, inpatient ward, medical or surgical intensive care unit after the patient has been assessed by the clinical team. If the primary diagnosis is septic shock, the clinical team will follow the hospital septic shock pathway. The diagnosis of septic shock as well as the type of the suspected infection will be left to the discretion of the patient's clinical team. Initial management according to the hospital septic shock pathway includes: giving IV fluids bolus, oxygen (if needed), and antibiotic based on the hospital antibiotic guidelines; and taking blood lactate, blood cultures, and other blood tests.
3. Recruitment and consent signing All patients who present to the study site's ED), inpatient ward, medical or surgical intensive care unit and diagnosed with septic shock will be approached for study participation. Each site will follow the Ministry of Public health in Qatar, MRC and the IRB guidelines regarding HIPAA authorization, informed consent and use of the Deferred Consent. Prior to obtaining consent or waiver, all potential subjects will undergo standard of care management procedures.

   The clinical team will obtain potential subject or legally authorized representative (LAR)/family agreement (verbally, but noted by ED, inpatient ward, MICU or SICU provider on screening form) to be approached by the study representative to participate. This will avoid "cold calling" coercion that could occur if direct contact by research team members was the initial method of assessing willingness to enroll. If that agreement is obtained, a trained study representative will approach the potential subject to gain written authorization and consent.

   In situations where the potential subject is unable to provide written authorization and consent, and their LAR/family is not available, it is permissible to use the Deferred Consent. Sites will seek this consent waiver according to the local standards and procedures.Detailed description of the recruitment and consent signing are available in the study protocol approved by the IRB
4. Randomization and initiation of study The investigators will assure that physicians (members of the study team) are available to prescribe the study interventions (triple therapy) in the ED, inpatient ward and the ICU, and will assure that required documentation of authorization and consent, or the Deferred Consent have been properly completed prior to enrollment in the study. Randomization will be 1:1 into each arm and will be done by computer via a web-based randomization system. If consent is refused, No data will be collected, as the IRB does not approve of any information collection for research from the patients if consent is not provided.

   The study investigator will inform the clinical team as soon as the treatment allocation is assigned. If the subject is assigned to the usual care, the clinical team will follow the hospital septic shock pathway. If the subject is assigned to the triple therapy arm, the clinical team will follow the hospital septic shock pathway plus the addition of the triple therapy as described previously in this protocol. The assigned clinical team will continue to provide all other aspects of care to the subject.
5. Study coordination and randomization details:

   Each study site will be led by a designated site coordinator. These individuals will attend the study training sessions at the Hamad General Hospital then they will in turn train physicians and nurses at their site to execute all relevant study procedures.

   The site coordinator will assure that study-trained physicians and nurses are available to perform the study interventions in the ED, inpatient ward and the ICU, and will be responsible to assure that study required documentation have been properly completed prior to enrollment in the study.

   Once the consent is obtained, inclusion criteria and other baseline data will be entered into a web-based enrollment application.

   Stratified block randomization will be used in the ratio of 1:1. Randomization will be stratified by study sites and will be done completely at random in order to conceal group allocation. Each enrolled subject will be assigned an identification number. If consent is refused, baseline characteristics will be collected to compare patients who did and did not enroll in the study to be used for analysis of potential selection bias and to determine the generalizability of the study results.

   Once a patient is allocated to triple therapy arm, the site coordinator will inform the clinical team and the intervention will begin in addition to other aspects of usual care
6. Study interventions

   1. Protocol delivery When a subject is assigned to the triple therapy, the study team receives a packet of the study materials. These will include an instruction sheet that outlines the protocol arm with accompanying data collection forms (flowsheet). A similar data collection form but without instructions or prompts, will be used by the site investigator for subjects in the 'usual care' arm to ensure equivalent data collection.

      If the subject is transferred from the ED or inpatient ward to the ICU and the protocol will continue as planned. At the end of the 7 days intervention, study medications will be discontinued to the extent possible.
   2. Data variables collected Study data in both arms will be collected by the unit study coordinator as per the study protocol, reviewed by the co-primary investigators, and will then become part of the subject's research record.
7. Adverse and disease-related events The research group will be responsible for notifying the DSMB regarding all reported AEs as per the definition and the procedures in the study protocol.
8. Data collection and statistical considerations Aim #1 and Aim #2: Mortality and Morbidity benefits:The primary hypotheses to be tested sequentially as part of Aim 1 are: Hypothesis 1, that triple therapy results in lower hospital mortality than usual care (arm A vs. arm B) and; Hypothesis 2, that that triple therapy results in lower hospital morbidity than usual care (arm A vs. arm B) The primary hypothesis to be tested as part of Aim 2 is that triple therapy results in no more adverse effects than placebo
9. Sample size We estimated that a total of 188 patients will give the study a power more than 80% to detect a relative risk reduction of approximately 50% in the primary outcome between the two arms assuming that the mortality in the control arm will be around 40% (based on institutional data and mortality rate in the control group of Marik study) using a two-sided test at significance level of 0.05.

   To be able to perform the interim analysis after recruitment of 50% of patients, the sample size is increased to 190 patients. We decided to enroll 212 patients (106 in each group) to account for 10% possible withdrawals.
10. Analysis plan The trial is designed to test the primary hypothesis (whether triple therapy is superior to usual care for treatment of septic shock).

    1. Descriptive analysis:

       Baseline characteristics and outcome data will be described as mean with standard deviation for continuous variables, median with interquartile range for ordinal variables and frequencies and percentages for categorical variables. The baseline characteristics will be compared between the two arms to observe balance and the success of randomization. These comparisons will not be subjected to statistical testing; as such tests are not recommended.
    2. Primary outcome: the number and percentage of hospital mortality after randomization will be reported for each treatment group. A multivariate logistic regression will be used with adjusted for APACHE II score at baseline. At the final analysis, the null hypothesis will be rejected when p<0.048. Analysis will be performed according to intention to treat principle.
11. Interim analysis is planned after recruitment of 50% of the predefined sample size (50 patients in each group). Decision to terminate the study at the interim analysis will be based on the O'Brien-Fleming boundary and will be taken by the DSMB as per the protocol. Thus, the study will be terminated if the two-sided P value of statistic test at the interim analysis is less than 0.005 and a boundary P value of 0.048 will be used for the statistical testing at the final analysis. If the intervention shows clinical superiority (defined as relative risk reduction of 10% or more) compared to usual care at the interim analysis but doesn't meet the statistical criteria for early termination, sample size adjustment will be performed. In this case, the sample size will be recalculated based on the observed event rates in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age (above 18 years old)
* Suspected or documented infection
* Meeting the definition of septic shock (Sepsis 3 definitions); Patients with septic shock can be identified with a clinical construct of sepsis with persisting hypotension requiring vasopressor therapy to maintain MAP ≥65 mm Hg and having a serum lactate level >2 mmol/L despite adequate volume resuscitation.
* Receiving norepinephrine at a dose equal or more than 0.1 µg/kg/min for more than or equal 6 hours.

Exclusion Criteria:

* Known pregnancy(1)
* Primary diagnosis of acute cerebral vascular event
* Acute coronary syndrome
* Status asthmaticus
* Major cardiac arrhythmia
* Active gastrointestinal hemorrhage
* Seizure
* Drug overdose
* Burn or trauma
* Requirement for immediate surgery(2)
* Absolute neutrophil count <500 mm3
* CD4 <50/mm³
* Do-not-resuscitate status
* Advanced directives restricting implementation of the protocol
* Terminally ill patients in palliative care
* Participation in another interventional study
* Known allergy or contraindication to one or more of the trial medications (Vitamin C, Thiamine, or Hydrocortisone)

  1. If the pregnancy status is unknown, the pregnancy test will not be done as part of the usual care, the patient is unconscious, and consent cannot be obtained for pregnancy test; we will not enroll the patient.
  2. Patients with septic shock and requiring immediate surgery will be evaluated after surgery for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-03-17 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Hospital Mortality at 60 days | 60 days after randomization
  Patients died during hospital admission

SECONDARY OUTCOMES:
Time to death | 60 days after randomization
  Time to death after randomization
Clinical evidence of organ dysfunction | 72 hours after randomization
  Change in SOFA* scores from admission to 72 hours
  *SOFA score is the Sequential Organ Failure Assessment score which is a mortality prediction score that is based on the degree of dysfunction of 6 organ systems. The score is made of 6 variables, each variable representing an organ system ( respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems). Each organ system score ranges from 0 (normal) to 4 (high degree of dysfunction/failure). The SOFA score ranges from 0 (normal) to 24 (high degree of dysfunction/failure)
Length of ICU stay | 60 days after randomization
  Duration the patient stayed in the ICU
Length of hospital stay | 60 days after randomization
  Duration the patient stayed in the hospital
Duration of vasopressor therapy | 60 days after randomization
  Time to discontinuation of vasopressor therapy and the MAP is more than 65 mmHg
Lactate clearance | 72 hours
  Defined as decrease in serum lactate levels over 72 hrs
Renal replacement therapy for acute kidney injury | 60 days after randomization
  Patient needed renal replacement therapy for acute kidney injury (Yes or no for each patient in both groups)
Need for Extracorporeal membrane oxygenation (ECMO) | 60 days after randomization
  Patient started on ECMO (Yes or no for each patient in both groups)

OTHER OUTCOMES:
Daily mean patient-day weighted blood glucose | 7 days after randomization
  Average of all blood glucose readings for a specific patient day then averaged across all patients of the arm.
Incidence of nephrolithiasis | 4 days after randomization
  Incidence of nephrolithiasis detected on radiological studies or diagnosed by the primary care team
Incidence of secondary infections | 60 days after randomization
  Incidence of secondary infections till ICU discharge
Mechanical ventilator weaning failure | 60 days after randomization
  Failure to pass a spontaneous breathing trial or the need for reintubation within 48 hours following extubation
Hypernatremia | 7 days after randomization
  serum sodium above 145 mEq/L
Hypokalemia | 7 days after randomization
  Serum potassium below 3.5 mEq/L
Hemolysis | 4 days after randomization
  Patient had hemolysis (Yes or no for each patient in both groups)
Gastrointestinal (GI) bleeding | 7 days after randomization
  Patient had GI bleeding (Yes or no for each patient in both groups)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelaty, MD, Principal Investigator — Hamad Medical Corporation; Adham Mohamed, PharmD, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martin GS, Mannino DM, Eaton S, Moss M. The epidemiology of sepsis in the United States from 1979 through 2000. N Engl J Med. 2003 Apr 17;348(16):1546-54. doi: 10.1056/NEJMoa022139. PMID 12700374
- [Result] Liu V, Escobar GJ, Greene JD, Soule J, Whippy A, Angus DC, Iwashyna TJ. Hospital deaths in patients with sepsis from 2 independent cohorts. JAMA. 2014 Jul 2;312(1):90-2. doi: 10.1001/jama.2014.5804. No abstract available. PMID 24838355
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Schorah CJ, Downing C, Piripitsi A, Gallivan L, Al-Hazaa AH, Sanderson MJ, Bodenham A. Total vitamin C, ascorbic acid, and dehydroascorbic acid concentrations in plasma of critically ill patients. Am J Clin Nutr. 1996 May;63(5):760-5. doi: 10.1093/ajcn/63.5.760. PMID 8615361
- [Result] Doise JM, Aho LS, Quenot JP, Guilland JC, Zeller M, Vergely C, Aube H, Blettery B, Rochette L. Plasma antioxidant status in septic critically ill patients: a decrease over time. Fundam Clin Pharmacol. 2008 Apr;22(2):203-9. doi: 10.1111/j.1472-8206.2008.00573.x. PMID 18353115
- [Result] Borrelli E, Roux-Lombard P, Grau GE, Girardin E, Ricou B, Dayer J, Suter PM. Plasma concentrations of cytokines, their soluble receptors, and antioxidant vitamins can predict the development of multiple organ failure in patients at risk. Crit Care Med. 1996 Mar;24(3):392-7. doi: 10.1097/00003246-199603000-00006. PMID 8625625
- [Result] Zabet MH, Mohammadi M, Ramezani M, Khalili H. Effect of high-dose Ascorbic acid on vasopressor's requirement in septic shock. J Res Pharm Pract. 2016 Apr-Jun;5(2):94-100. doi: 10.4103/2279-042X.179569. PMID 27162802
- [Result] Tanaka H, Matsuda T, Miyagantani Y, Yukioka T, Matsuda H, Shimazaki S. Reduction of resuscitation fluid volumes in severely burned patients using ascorbic acid administration: a randomized, prospective study. Arch Surg. 2000 Mar;135(3):326-31. doi: 10.1001/archsurg.135.3.326. PMID 10722036
- [Result] Nathens AB, Neff MJ, Jurkovich GJ, Klotz P, Farver K, Ruzinski JT, Radella F, Garcia I, Maier RV. Randomized, prospective trial of antioxidant supplementation in critically ill surgical patients. Ann Surg. 2002 Dec;236(6):814-22. doi: 10.1097/00000658-200212000-00014. PMID 12454520
- [Result] Fowler AA 3rd, Syed AA, Knowlson S, Sculthorpe R, Farthing D, DeWilde C, Farthing CA, Larus TL, Martin E, Brophy DF, Gupta S; Medical Respiratory Intensive Care Unit Nursing; Fisher BJ, Natarajan R. Phase I safety trial of intravenous ascorbic acid in patients with severe sepsis. J Transl Med. 2014 Jan 31;12:32. doi: 10.1186/1479-5876-12-32. PMID 24484547
- [Result] Donnino MW, Carney E, Cocchi MN, Barbash I, Chase M, Joyce N, Chou PP, Ngo L. Thiamine deficiency in critically ill patients with sepsis. J Crit Care. 2010 Dec;25(4):576-81. doi: 10.1016/j.jcrc.2010.03.003. Epub 2010 Jun 19. PMID 20646908
- [Result] Donnino MW, Andersen LW, Chase M, Berg KM, Tidswell M, Giberson T, Wolfe R, Moskowitz A, Smithline H, Ngo L, Cocchi MN; Center for Resuscitation Science Research Group. Randomized, Double-Blind, Placebo-Controlled Trial of Thiamine as a Metabolic Resuscitator in Septic Shock: A Pilot Study. Crit Care Med. 2016 Feb;44(2):360-7. doi: 10.1097/CCM.0000000000001572. PMID 26771781
- [Result] Marik PE, Zaloga GP. Adrenal insufficiency during septic shock. Crit Care Med. 2003 Jan;31(1):141-5. doi: 10.1097/00003246-200301000-00022. PMID 12545007
- [Result] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Crit Care Med. 2017 Mar;45(3):486-552. doi: 10.1097/CCM.0000000000002255. PMID 28098591
- [Result] Keh D, Trips E, Marx G, Wirtz SP, Abduljawwad E, Bercker S, Bogatsch H, Briegel J, Engel C, Gerlach H, Goldmann A, Kuhn SO, Huter L, Meier-Hellmann A, Nierhaus A, Kluge S, Lehmke J, Loeffler M, Oppert M, Resener K, Schadler D, Schuerholz T, Simon P, Weiler N, Weyland A, Reinhart K, Brunkhorst FM; SepNet-Critical Care Trials Group. Effect of Hydrocortisone on Development of Shock Among Patients With Severe Sepsis: The HYPRESS Randomized Clinical Trial. JAMA. 2016 Nov 1;316(17):1775-1785. doi: 10.1001/jama.2016.14799. PMID 27695824
- [Result] Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. Chest. 2017 Jun;151(6):1229-1238. doi: 10.1016/j.chest.2016.11.036. Epub 2016 Dec 6. PMID 27940189
- [Result] Fujita I, Hirano J, Itoh N, Nakanishi T, Tanaka K. Dexamethasone induces sodium-dependant vitamin C transporter in a mouse osteoblastic cell line MC3T3-E1. Br J Nutr. 2001 Aug;86(2):145-9. doi: 10.1079/bjn2001406. PMID 11502226
- [Result] Annane D, Timsit JF, Megarbane B, Martin C, Misset B, Mourvillier B, Siami S, Chagnon JL, Constantin JM, Petitpas F, Souweine B, Amathieu R, Forceville X, Charpentier C, Tesniere A, Chastre J, Bohe J, Colin G, Cariou A, Renault A, Brun-Buisson C, Bellissant E; APROCCHSS Trial Investigators. Recombinant human activated protein C for adults with septic shock: a randomized controlled trial. Am J Respir Crit Care Med. 2013 May 15;187(10):1091-7. doi: 10.1164/rccm.201211-2020OC. PMID 23525934
- [Result] Campbell GD Jr, Steinberg MH, Bower JD. Letter: Ascorbic acid-induced hemolysis in G-6-PD deficiency. Ann Intern Med. 1975 Jun;82(6):810. doi: 10.7326/0003-4819-82-6-810_1. No abstract available. PMID 1138591
- [Result] Campbell A, Jack T. Acute reactions to mega ascorbic acid therapy in malignant disease. Scott Med J. 1979 Apr;24(2):151-3. doi: 10.1177/003693307902400210. PMID 227054
- [Result] Riordan HD, Casciari JJ, Gonzalez MJ, Riordan NH, Miranda-Massari JR, Taylor P, Jackson JA. A pilot clinical study of continuous intravenous ascorbate in terminal cancer patients. P R Health Sci J. 2005 Dec;24(4):269-76. PMID 16570523
- [Result] Deyo RA, Cherkin DC, Ciol MA. Adapting a clinical comorbidity index for use with ICD-9-CM administrative databases. J Clin Epidemiol. 1992 Jun;45(6):613-9. doi: 10.1016/0895-4356(92)90133-8. PMID 1607900
- [Result] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Result] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Derived] Mohamed A, Abdelaty M, Saad MO, Shible A, Mitwally H, Akkari AR, Elbuzidi A, Bintaher A, Hashim A, Abdelrahim M, Afzal M, El-Enany R, El-Hamid M, Bakdach D, Karic E, Shehatta A, Ibrahim AS, Lance M, Hssain AA, Hassan I. EVALUATION OF HYDROCORTISONE, VITAMIN C, AND THIAMINE FOR THE TREATMENT OF SEPTIC SHOCK: A RANDOMIZED CONTROLLED TRIAL (THE HYVITS TRIAL). Shock. 2023 May 1;59(5):697-701. doi: 10.1097/SHK.0000000000002110. Epub 2023 Mar 8. PMID 36870070